CLINICAL TRIAL: NCT02606318
Title: Adjusting Challenge-Skill Balance to Improve the Elderly's Quality of Life: A Randomized Controlled Trial
Brief Title: Adjusting Challenge-Skill Balance to Improve the Elderly's Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harue Hospital (Other)
Responsible Party: Principal Investigator, Ippei Yoshida, MS, OTR, Harue Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YIPPE-1
Record Dates: First submitted 2015-11-07; First posted 2015-11-17 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Elderly
Keywords: Occupational Therapy; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjusted the challenge-skill balance (Experimental): This group received 10-session occupational therapy with adjustment of challenge-skill balance.This intervention aimed at improving the skill level for the activity has started once the balance were balanced.
  Interventions: Other: Adjusted the challenge-skill balance
- Non-adjusted the challenge-skill balance (Other): This group received 10-session occupational therapy without adjustment of challenge-skill balance. That is conducted the therapy in the normal manner for the day care center.
  Interventions: Other: Non-adjusted the challenge-skill balance

INTERVENTIONS:
Other: Adjusted the challenge-skill balance — In the first session of occupational therapy, the therapist assessed the client's problems in daily living using the Canadian Occupational Performance Measure. Based on the problems identified, an activity that could be supported in day care was selected. In the second session, the client performed the selected activity, and then the challenge and skill levels of the activity were evaluated. Based on these levels, adjustment of the challenge-skill balance in the activity was attempted. Occupational therapy consisted of 10 sessions of 20 minutes held over about 10 weeks
  Arms: Adjusted the challenge-skill balance
Other: Non-adjusted the challenge-skill balance — The first and second sessions were conducted in the same way as for the experimental group, except that the therapists were not informed of the client's subjective perception of the challenge and skill levels for the activity. From the third session, the therapists simply assessed the client's performance and conducted the therapy in the normal manner for the day care center, following the general guidelines for occupational therapy practice
  Arms: Non-adjusted the challenge-skill balance

SUMMARY:
The purpose of this study was to clarify the effects on health-related QOL of occupational therapy involving the adjustment of challenge-skill balance in the activity of elderly clients.

DETAILED DESCRIPTION:
This study was single-blind, randomized controlled trial. Clients were randomly assigned by blocked randomization (block size 4) to either the experimental group (occupational therapy that included assessment and adjustment of the challenge-skill balance of the activities) or to the control group (occupational therapy as normally conducted at the day care center). Randomization was stratified by sex and EuroQol visual analogue scale, resulting in four layers. The primary outcome was change in health-related quality of life after 10 sessions of occupational therapy. Clients were assessed before the intervention (pre-test) and after the 10th session (post-test). Significant differences were observed in the EuroQol-5 Dimension (EQ-5D) score and in the Medical Outcome Study 8-Item Short-Form Health Survey (SF-8) scores for general health, physical functioning , and vitality.

ELIGIBILITY:
Inclusion Criteria:

* age >60 years
* occupational therapy at the center for >3 months

Exclusion Criteria:

* dementia
* visual impairment

Ages: 62 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in the EuroQol-5 Dimension questionnaire | Baseline and 10 weeks
  The EQ-5D defines health in five dimensions (mobility, self-care, usual activities, pain and discomfort, and anxiety or depression). The EQ-5D also has a visual analogue scale (EQ-VAS) that enables self-assessment on a scale from 0 (worst possible health) to 100 (best possible health).
Change in the Medical Outcome Study 8-Item Short-Form Health Survey questionnaire | Baseline and 10 weeks
  The SF-8 encompasses eight domains: general health, physical functioning, role physical, bodily pain, vitality, social functioning, role emotional, and mental health, which can be combined to yield a physical component summary score and a mental component summary score.

SECONDARY OUTCOMES:
Change in the Flow State Scale for Occupational Tasks questionnaire | Baseline and 10 weeks
  Flow State Scale for Occupational Tasks is a scale that can measure a patient's flow state in a clinical situation such as occupational therapy
Change in the Canadian Occupational Performance Measure questionnaire | Baseline and 10 weeks
  Canadian Occupational Performance Measure assesses client's self-perception of their occupational performance

CONTACTS AND LOCATIONS:
Overall Officials: Tetsushi Nonaka, Ph.D, Principal Investigator — Graduate School of Human Development and Environment

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Hirao K, Kobayashi R, Okishima K, Tomokuni Y. Flow experience and health-related quality of life in community dwelling elderly Japanese. Nurs Health Sci. 2012 Mar;14(1):52-7. doi: 10.1111/j.1442-2018.2011.00663.x. Epub 2012 Jan 30. PMID 22288733